CLINICAL TRIAL: NCT05365672
Title: An Open, Randomized-controlled, Multi-center Phase-II Clinical Trial of Individualized Immunosuppression With Intravenously Administered Donor Modified Immune Cells (MIC) Compared to Standard-of-care in Living Donor Kidney Transplantation
Brief Title: Clinical Trial With Donor Modified Immune Cells in Living Donor Kidney Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TolerogenixX GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOL-2
Record Dates: First submitted 2022-04-26; First posted 2022-05-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Kidney Transplantation
Keywords: living donor kidney transplantation; TOL-2; modified immune cells; MIC; mitomycin C; peripheral blood mononuclear cells; PBMC; kidney donor; TolerogenixX; tolerance; immunosuppression; donor-specific unresponsiveness; EudraCT No. 2021-000561-33
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MIC with low immunosuppression (Experimental): Patients in MIC Arm A receive the investigational medicinal product MIC plus immunosuppression consisting of tacrolimus, mycophenolic acid derivative and corticosteroids (without IL-2 receptor antibody induction therapy).
  Tacrolimus dose will be gradually reduced to 4-8 μg/L at Day 183 and the corticosteroid treatment will be stopped at Day 92 after gradual dose reduction.
  Interventions: Biological: MIC
- MIC with minimal immunosuppression (Experimental): Patients in MIC Arm B receive the investigational medicinal product MIC plus immunosuppression consisting of tacrolimus, mycophenolic acid derivative and corticosteroids (without IL-2 receptor antibody induction therapy).
  Tacrolimus dose will be gradually reduced to 4-8 μg/L at Day 183 and the corticosteroid treatment will be stopped at Day 92 after gradual dose reduction.
  The mycophenolic acid derivative will be stopped between Days 141 and 182.
  Interventions: Biological: MIC
- Standard of care immunosuppression for transplantation (Other): Patients of the Control Arm receive standard of care immunosuppression for kidney transplantations according to the Efficacy Limiting Toxicity Elimination (ELITE) symphony scheme (interleukin [IL]-2 receptor antibody induction therapy, tacrolimus, mycophenolic acid derivative and corticosteroids) without the investigational medicinal product MIC.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: MIC — Single intravenous infusion of 1.5x10exp8 MIC per kg of body weight
  Arms: MIC with low immunosuppression; MIC with minimal immunosuppression
Other: Standard of Care — No application of the investigational medicinal product MIC
  Arms: Standard of care immunosuppression for transplantation

SUMMARY:
In this clinical trial the investigational medicinal product MIC is to be examined for its efficacy and safety in patients with living kidney transplantation. For this purpose the patients participating in the clinical trial and their associated kidney donors are randomly assigned to one of three treatment groups during the screening procedure. For the production of the investigational medicinal product MIC for the patients in the MIC therapy group mononuclear cells of the peripheral blood are obtained from the donors in a leukapheresis procedure. In the subsequent treatment phase, the patients in the MIC therapy group receive MIC as a weight-adjusted single dose administered intravenously. As part of the 12-month follow-up phase the kidney transplant and the corresponding immunosuppressive therapy will take place seven days later. Patients in the control group will receive a conventional standard immunosuppressive regimen without prior administration of the investigational medicinal product MIC after kidney transplantation. All patients taking part in this clinical trial are followed up for one year after kidney transplantation with regard to the efficacy and safety of MIC in regular visits at their study site. As the investigational medicinal product is an advanced therapy medicinal product (ATMP) all subjects will be monitored for a further 2 years after the end of the follow-up phase of the clinical trial.

A total of 63 transplant pairs, consisting of donor and transplant recipient, are to be included in the clinical trial. The 63 patients will be randomized 2:1 to be treated with MIC (MIC group) or without MIC (control group). Additionally, low immunosuppression or minimal immunosuppression treatments will be used in the patients in the MIC group.

ELIGIBILITY:
Inclusion Criteria:

Donors:

1. Age ≥18 years and able to consent
2. Ability to understand the nature and scope of the clinical trial
3. Written consent form given prior to any trial-related procedures (including PBMC donation)

Patients:

1. Patient with CKD in stage 5 (e.g., estimated glomerular filtration rate [eGFR] <15 mL/min and/or on renal replacement therapy), who are in preparation for kidney transplantation from a live donor
2. Age ≥18 years, <70 years
3. ABO-blood group identical or compatible with donor
4. First kidney transplantation
5. Complement dependent cytotoxicity (CDC)-panel reactive antibodies <20%
6. No detection of a donor-specific HLA-antibody in the Luminex-Assay (cutoff: mean fluorescence intensity [MFI] ≤1,000)
7. Negative CDC crossmatch with the donor
8. Negative PCR test result for severe acute respiratory syndrome coronavirus-2 (SARSCoV-2) at Screening
9. Patient's living donor gave written consent for trial participation
10. Ability to understand the nature and scope of the clinical trial
11. Written informed consent given prior to any trial-related procedures
12. Female patients of childbearing potential must:

    1. have a negative pregnancy test (blood) at Screening.
    2. either commit to true abstinence from heterosexual contact or agree to use, and be able to comply with, 2 highly effective measures of contraception control (failure rate less than 1% per year when used consistently and correctly) without interruption, during the trial participation. Patients who discontinue mycophenolic acid derivate during the trial participation can switch to 1 highly effective contraceptive method 6 weeks after the end of mycophenolic acid derivative treatment. Reliable methods for this trial are: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone releasing system, bilateral tubal occlusion, sexual abstinence or vasectomized sexual partner. Abstinence from heterosexual contact is only accepted as true abstinence: when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods and withdrawal] is not an acceptable method of contraception.) Postmenopausal (no menses for at least 1 year without alternative medical cause) or surgically sterile female patients (tubal ligation, hysterectomy or bilateral oophorectomy) may be enrolled.
    3. agree to abstain from breast feeding during the trial participation.
13. Male patients must practice true abstinence or agree to use a condom during sexual contact with a pregnant woman or a woman of childbearing potential during the trial participation and for at least 90 days after the end of mycophenolic acid derivative treatment, even if he has undergone a successful vasectomy.

Exclusion Criteria:

Donors:

1. Pregnant or breastfeeding
2. Participation in an interventional clinical trial within 30 days prior to Screening or in observation period of a competing study
3. Severe psychiatric disease
4. Severe cardiovascular diseases (i.e., heart insufficiency of grade NYHA III or IV)
5. Severe neurological diseases
6. Severe liver or kidney diseases
7. Any acute or chronic disease that may put the donor at risk in case of cell donation by leukapheresis
8. Malignant neoplasms, except in situ carcinoma after complete removal
9. Known infections or exposures to human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), hepatitis E virus, West Nile virus (WNV; testing only required during WNV season [June 1st to November 30th of a year]), gonorrhea or syphilis, with the risk of transmission of infection (Note: If tested positive for EBV immunoglobulin [Ig]M, an EBV PCR test has to be performed for confirmation)
10. Active bacterial, mycotic or viral infection, except active infections that, in the investigator's opinion, do not affect patient safety (e.g., foot fungus, nail fungus, or common warts)
11. Known malaria infection; known infection of tuberculosis, Q fever, Salmonella typhi and paratyphi, or osteomyelitis (if not medically documented to have been cured for 2 years); known toxoplasmosis (except if symptom free for 6 months); after completion of treatment for rheumatic fever (except if treatment was completed for 2 years)
12. Known transmissible spongiform encephalopathies
13. Known protozoonosis (babesiosis, trypanosomiasis [e.g., chagas], leishmaniosis), known chronic bacterial infections as brucellosis, rickettsiosis, leprosy, relapsing fever, melioidosis, tularemia (except after assured healing according to documented medical assessment)
14. Autoimmune diseases requiring systemic immunosuppressive therapy
15. Allergies requiring systemic immunosuppressive therapy
16. Immunosuppressive therapy within 6 months prior screening
17. Known or suspected abuse of alcohol, drugs, or medicinal products
18. Unexplained night sweats, unexplained fever, unexplained weight loss, prolonged unexplained cough or diarrhea, unexplained skin lesions, lymph gland swelling or thrush
19. Dura mater and/or cornea grafts, allogeneic organ transplants, xenotransplants, pituitary hormones of human origin received
20. Stay of longer than 6 months in the United Kingdom between 1980 and 1996 and/or an operation and/or blood transfusion in the United Kingdom after 01-Jan-1980
21. Operations or other invasive interventions (e.g., endoscopies, biopsies, catheter applications, acupunctures [except acupuncture with sterile and/or disposable needles]) within 4 months prior to Screening
22. Any invasive exposure to blood (i.e., allogeneic blood components or plasma derivatives) or blood-contaminated injection needles or instruments, tattoos or piercings within 4 months prior to Screening
23. Positive PCR test result for SARS-CoV-2 at Screening
24. Hemoglobin <8.0 g/dL, thrombocytes <80,000/μL and/or leukocytes <3,000/μL
25. Known history of hypersensitivity to components used in the leukapheresis setting (i.e., components of the anticoagulant acid citrate dextrose solution)
26. Any finding or medical condition prohibiting the inclusion in the trial according to the judgment of the responsible leukapheresis physician (including assessment of the suitability of the veins for leukapheresis by the investigator)

Patients:

1. Preexisting severe psychiatric disorder
2. Heart insufficiency of grade NYHA III or IV
3. Severe liver disease (aspartate aminotransferase or alanine aminotransferase or gamma glutamyl transpeptidase ≥3 x ULN)
4. Active infection of HIV, HBV, HCV, EBV or syphilis
5. Active bacterial, mycotic, or viral infection, except active infections that, in the investigator's opinion, do not affect patient safety (e.g., foot fungus, nail fungus, or common warts)
6. Negative serological test result for antibodies specific for Epstein-Barr virus (EBV) antigens (Note: EBV negative patients can be included if the donor is confirmed EBV negative)
7. Malignant disease within 2 years prior to Screening, except basal cell carcinomas of the skin and in situ carcinomas
8. Immunosuppressive therapy (e.g., for the treatment of an auto-immune disease) within 6 months prior Screening
9. Preexisting vasculitis or collagenosis
10. Known presence of irregular antibodies in Coombs test
11. Vaccination within 4 weeks prior to Screening
12. Spleen removed
13. Known or suspected abuse of alcohol, drugs, or medicinal products
14. Pregnant or breastfeeding
15. Female patients who have a child with the donor or were pregnant from the donor due to possible sensitization
16. Known history of hypersensitivity to the cellular components or to any other constituent/excipient in the pharmaceutical formulation of MIC (e.g., components of the SSP+ buffer as electrolytes (sodium chloride, potassium chloride, magnesium), citrate and phosphate, traces of mitomycin C, human albumin, or EDTA)
17. Any finding or medical condition prohibiting the inclusion in the trial according to the judgment of the investigator
18. Participation in an interventional clinical trial within 30 days prior to Screening or in observation period of a competing study
19. Employees of the sponsor, or employees or relatives of the investigator

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
No acute rejection, graft loss, graft dysfunction | On day 367 post investigational medicinal product application
  Proportion of patients who achieve an operational tolerance-like phenotype compared to standard of care therapy defined on Visit Day 367 as fulfilling four criteria that are evaluated:
  Criterium 1.: No acute rejection (biopsy-proven as >Banff Borderline or clinically suspected rejection according to evaluation of adjudication committee), graft loss, graft dysfunction (eGFR <30 mL/min), or death on Visit Day 367
No development of de novo donor-specific HLA- antibodies | Between day 0 and day 367 post investigational medicinal product application
  Proportion of patients who achieve an operational tolerance-like phenotype compared to standard of care therapy defined on Visit Day 367 as fulfilling four criteria that are evaluated:
  Criterium 2.: No development of donor-specific HLA antibodies (DSA ≤1,000 MFI; values >1,000 MFI after Visit Day 6 has to be confirmed by second measurement after 4 weeks) until Visit Day 367 as measured by Luminex single antigen test
Induction of regulatory B cells (Breg) to ≥3% | On day 367 post investigational medicinal product application
  Proportion of patients who achieve an operational tolerance-like phenotype compared to standard of care therapy defined on Visit Day 367 as fulfilling four criteria that are evaluated:
  Criterium 3.: Induction of Breg ≥3% measured on Visit Day 367 (patient has to be infection-free at timepoint of measurement)
Patient on tacrolimus therapy with ≤720 mg EC-MPS and no corticosteroids | Between days 277 and 367 post investigational medicinal product application
  Proportion of patients who achieve an operational tolerance-like phenotype compared to standard of care therapy defined on Visit Day 367 as fulfilling four criteria that are evaluated:
  Criterium 4.: Patient on tacrolimus therapy with ≤720 mg EC-MPS and no corticosteroids (as well as no other immunosuppressive drug) on Visit Day 277 and remaining on this therapy until Visit Day 367

SECONDARY OUTCOMES:
Key secondary: Number of patient-relevant infections during the first year after transplantation | On day 367 post investigational medicinal product application
  Safety evaluation of MIC treatment versus standard of care therapy is based on number of patient-relevant infections during the first year after transplantation.
  Patient-relevant infections are:
  Pneumonia, and/or complicated urinary tract infection, and/or sepsis from any cause, and/or opportunistic infection.
Key secondary: Biopsy proven acute rejection, graft loss, graft dysfunction, or death | On day 367 post investigational medicinal product application
  Safety evaluation of MIC treatment versus standard of care therapy is also based on proportion of patients with acute rejection (biopsy-proven as >Banff Borderline or clinically suspected rejection according to evaluation of adjudication committee), graft loss, graft dysfunction, or death on Visit Day 367
Number of Adverse Events (AEs) including serious AEs and AEs of special interest | From screening through study completion, 3 years estimated.
  Determine safety and efficacy of MIC treatment based on AE outcome
Frequency of local or systemic reactions as result of MIC application | From day 0 through study completion, 3 years estimated.
  Determine safety and efficacy of MIC treatment based on further parameters other than comparison to standard of care therapy
Monitoring of patient survival | On Visit Days 187 and 367 post investigational medicinal product application
  Determine safety and efficacy of MIC treatment based on further parameters other than comparison to standard of care therapy: Monitoring for death of patient.
Monitoring of graft kidney survival | On Visit days 187 and 367 post investigational medicinal product application
  Determine safety and efficacy of MIC treatment based on further parameters other than comparison to standard of care therapy: Monitoring for death of grafted kidney.
Incidence of biopsy-proven acute rejections and time to first rejection (>Banff Borderline) | On Visit Days 97 and 142 post investigational medicinal product application
  Assessment is done according to current version Banff criteria and confirmed by a blinded central pathologist
Molecular scores in molecular microscope diagnostic system (MMDx) | On Visit Day 367 post investigational medicinal product application
  Molecular biopsy analysis using MMDx will be done
Percentage of patients who achieved tacrolimus and EC-MPS dual therapy or tacrolimus monotherapy | On day 367 post investigational medicinal product application
  Percentage of patients who achieved tacrolimus and EC-MPS dual therapy in the MIC Arm A or Control Arm or tacrolimus monotherapy in the MIC Arm B
Amount of donor-specific HLA antibodies (DSA) | On Visit Days 6, 187 and 367 post investigational medicinal product application
  DSA measurement (>1,000 MFI; confirmed by second measurement after 4 weeks for assessments after Day 6) will be done by blinded Luminex single antigen test
Occurrence of delayed function of the kidney graft after transplantation | On Visit Day 37 post investigational medicinal product application
  Defined as dialysis within the first week after transplantation, except for one dialysis for hyperkalemia
Assessment of estimated Glomerular Filtration Rate (eGFR) [CKD-EPI]) | From screening through study completion, 3 years estimated.
  Measurement of eGFR according to chronic kidney disease epidemiology collaboration (CKD-EPI)
Assessment of the incidence of cytomegalovirus (CMV) reactivation (CMV-DNA ≥1,000 copies/mL) | From screening through study completion, 3 years estimated.
  CMV amount will be measured as CMV-DNA copies/mL
Assessment of the incidence of BK virus replication ≥10,000 copies/mL | From screening through study completion, 3 years estimated.
  BK virus amount will be measured as DNA copies/mL
Assessment of the incidence of BK virus associated nephropathy | From screening through study completion, 3 years estimated.
  Nephropathy will be assessed using biopsy material
Assessment of the incidence of hospital readmissions after transplant surgery | On days 5, 7, 37, 97, 142, 187, 277, 367, month 24, 36 post investigational medicinal product application
  Assessment of the number of patients who had hospital readmissions after transplant surgery
Assessment of days in hospital, on intensive care and hours on mechanical ventilation upon re-admission | On day -14 to -7 and 367 post investigational medicinal product application
  Assessment of days in hospital, on intensive care and hours on mechanical ventilation (the treatment to help a person breathe when they find it difficult or are unable to breathe on their own) that patients needed upon hospital re-admission after transplant surgery
Change in quality of life as assessed by questionnaire | Between day -14 to -7 and 367 post investigational medicinal product application
  The SF-36 questionnaire with 36 questions will be used to assess the change in quality of life between screening and first year after treatment
Incidence of new-onset diabetes mellitus after transplantation | From day 0 through study completion, 3 years estimated.
  Assessment of incidence of diabetes mellitus after transplantation by measuring fasting plasma glucose (≥7.0 mmol/L / 126 mg/dL) with no calorie intake for at least 8 hours
Determination of therapeutic intensity score (TIS) based on blood pressure on Visit Day 367 compared to Baseline | On day -14 to -7 and 367 post investigational medicinal product application
  Assessment of the TIS as a summary measure that accounts for the number and the relative doses of blood pressure medications for a patient by a blinded adjudication committee one year after treatment
Breg percentage | On day 367 post investigational medicinal product application
  Assessment of the percentage of regulatory B cells of the white blood cell population measured from blood samples by Fluorecscence Activated Cell Sorting (FACS)
Anti-donor T cell response to the donor | From day 0 through study completion, 3 years estimated.
  Anti-donor T cell response will be assessed from blood samples using the mixed lymphocyte reaction in vitro assay
Cumulative steroid dose during the first year after treatment | On day 367 post investigational medicinal product application
  Assessment of the overall amount of steroids given to the patient as immunosuppressive treatment during the first year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Christian Morath, Prof.Dr.med., Principal Investigator — University Hospital Heidelberg
Locations (8):
- Germany (8):
  - Medizinische Klinik mit Schwerpunkt Nephrologie und Internistische Intensivmedizin Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Universitäres Transplantations Centrum, Hamburg
  - Innere Medizin V; Klinik für Hämatologie, Onkologie, Rheumatologie; Universitätsklinikum Heidelberg, Heidelberg
  - Medizinische Klinik, Innere Medizin X Nephrologie - Nierenzentrum Universitätsklinikum Heidelberg, Heidelberg
  - Transplantationszentrum München; Ludwig-Maximilians-Universität, Munich
  - Klinikum rechts der Isar, Abteilung Nephrologie, Technische Universität München, Munich
  - Universitätsklinikum Münster, Transplantationsnephrologie, Münster
  - Klinik für Nieren-, Hochdruck- und Autoimmunerkrankungen; Transplantationszentrum Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morath C, Schmitt A, Schmitt M, Wang L, Kleist C, Opelz G, Susal C, Tran TH, Scherer S, Schwenger V, Kemmner S, Fischereder M, Stangl M, Hauser IA, Sommerer C, Nusshag C, Kalble F, Speer C, Benning L, Bischofs C, Sauer S, Schubert ML, Kunz A, Huckelhoven-Krauss A, Neuber B, Mehrabi A, Schwab C, Waldherr R, Sander A, Busch C, Czock D, Bohmig GA, Reiser J, Roers A, Muller-Tidow C, Terness P, Zeier M, Daniel V, Schaier M. Individualised immunosuppression with intravenously administered donor-derived modified immune cells compared with standard of care in living donor kidney transplantation (TOL-2 Study): protocol for a multicentre, open-label, phase II, randomised controlled trial. BMJ Open. 2022 Nov 11;12(11):e066128. doi: 10.1136/bmjopen-2022-066128. PMID 36368749